# School Water Access, Food and Beverage Intake, and Obesity Informed Consent Form

NCT03181971

February 29, 2024

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

| FOR QUESTIONS ABOUT THE STUDY, CONTACT: | Dr. | , at |
|-----------------------------------------|----------|------|
| , or by I | phone at | |

**DESCRIPTION:** Your child is invited to participate in a research study on how promoting drinking water in schools impacts what students eat and drink, and also their growth.

Drinking water can help children learn, maintain a healthy weight, and prevent cavities. Yet at many schools, students have limited access to water during the school day.

Your child's school has agreed to participate in this study, which includes the following activities to promote intake of water:

- Installation of safe and appealing water fountains and water bottle filling stations at the school
- Educational school assembly about the importance of drinking water
- Eight short lessons for 4<sup>th</sup> graders about why drinking water is important. Each 4<sup>th</sup> grade student will also receive two free Bisphenol A (BPA)-free reusable water bottles for use at home and at school and other small prizes

Additionally, your child's school principal has agreed to allow researchers to conduct evaluation activities to understand how the project impacts what students eat and drink and also their growth. Your child will be asked to:

- Allow researchers to visit the school to observe what students drink at school
- Allow Dr. and her research team to complete height and weight measurements. Dr. and her research team will use standard techniques outlined by the National Health and Nutrition Examination Survey Anthropometry Procedures Manual. Height and weight measurements are similar to how your child is measured at the doctor's office and in schools in 5th, 7th, and 9th grade. Measurements of students will occur one at a time and will take place in a private area. Students will only be asked to remove heavy coats and shoes for the measurements. We will take these measurements three times -- once now, once again before the end of the school year and once more during the next school year.
- Participate in short surveys. At the same time as the height and weight measurements, your child will be asked to complete a short survey with questions about beverage intake, screen time, and physical activity.
- Complete food and beverage diaries. Researchers will teach your child's class how to fill
  out a 24-hour diary to record all the food and beverages they consume in one day. Your
  child will be asked to complete the diary at home with your help two times -- once now
  and once again before the end of the school year.

The National Institutes of Health is providing financial support and/or material for this study.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

**RISKS AND BENEFITS:** The risks associated with this study are minimal and include the possibility (1) that your child may feel uncomfortable while being measured and weighed and (2) loss of privacy. We will ensure that all height and weight measurements are collected quietly and in a private area. We will also do our best to protect the information we collect from your child. Information that identifies your child will be kept secure. The height and weight measurements and food and beverage diaries will not include details that directly identify your child, such as your child's name or address. Only a small number of researchers will have direct access to the information. Any reports from the study will not mention individual children or schools.

Another possible risk is that underweight children could lose weight as a result of this study. If your child is considered to be underweight (their Body Mass Index or BMI is in the fifth percentile or lower), will contact you to discuss strategies for healthy weight management.

We cannot and do not guarantee or promise that your child will receive any benefits from this study. However, the information that your child provides may help schools, public health officials, policymakers to better understand how improvements in water access and promotion affects what students eat and drink, and their health. Your child is free to not participate in the study. If you decide not to allow your child to take part in this study, there will be no penalty to you or your child, and your child's relationship with his/her school or Stanford University will not be impacted in any way.

**TIME INVOLVEMENT:** Your child's participation in this study will take approximately 5 hours total over the course of the 18 month study.

**PAYMENTS:** Your child will receive a \$10 movie theater gift card after turning in all food and beverage diaries and surveys for his/her participation. Students will also receive reusable water bottles and small prizes during lessons and for completing home activities during the study.

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to allow your child to participate in this project, please understand your child's participation is voluntary and you have the right to withdraw your consent or discontinue your child's participation at any time without penalty or loss of benefits to which you are otherwise entitled. The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your child's identity will not be disclosed. Your child has the right to refuse to answer particular questions.

**CERTIFICATE OF CONFIDENTIALITY:** This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

It is possible that, based on information gained from this study, the researchers may have serious concerns (relating to matters such as severe depression, physical abuse, etc.) about your child's health and/or safety; in such a case, the researchers may contact you and provide a referral for your child's care. It is possible that, based on information gained from this study, the researchers may be required to report information (e.g., information relating to suicide, physical or sexual abuse) to the appropriate authorities.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## **Authorization To Use Your Child's Health Information For Research Purposes**

Because information about your child and your child's health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your child's health information will be used or disclosed in the study. Your child's information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my child's health information be utilized in the study?

This is a research study to investigate how promoting drinking water in schools impacts what students eat and drink, and their growth. The information that your child provides may help schools, public health officials, and policymakers to better understand how promoting water in schools can affect students' health. The results of this research study may be presented at scientific meetings, published in scientific journals, or provided in reports to the funding agency, the National Institutes of Health. However, your child's identity and your child's school name will not be disclosed.

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, your child will not be able to participate in this research study. Signing the form is not a condition for receiving any medical care outside of the study.

## If I sign, can I revoke it or withdraw from the research later?

If you allow your child to participate, you are free to withdraw your authorization regarding the use and disclosure of your child's health information (and to discontinue any other participation in the study) at any time. After any revocation, your child's health information will no longer be used or disclosed in the study, except to the extent that the law allows us to continue using your child's information (e.g., necessary to maintain integrity of research). If you wish to revoke your authorization for the research use or disclosure of your child's health information in this study, you must write to:

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## What Personal Information Will Be Obtained, Used or Disclosed?

Your child's health information related to this study name, date of birth, height/weight, and beverage and food intake may be used or disclosed in connection with this research study.

## Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your child's health information in connection with this research study:

- The Protocol Director, Dr.
- The Stanford University Administrative Panel on Human Subjects in Medical Research and any other unit of Stanford University as necessary
- Research Staff

## Who May Receive or Use the Information?

The parties listed in the preceding paragraph may disclose your child's health information to the following persons and organizations for their use in connection with this research study:

- The Office for Human Research Protections in the U.S. Department of Health and Human Services
- National Institutes of Health

Your child's information may be re-disclosed by the recipients described above, if they are not required by law to protect the privacy of the information.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## When will my authorization expire?

Your authorization for the use and/or disclosure of your child's health information will end on May 31, 2030 or when the research project ends, whichever is earlier.

| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |
|---|---|
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g., parent, guardian or conservator) | |

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and

| Obesity | |
|---|---|
| and the research team may also withdraw you consent for one or more of the following reasons: Failure to follow the instructions of Dr. Dr. decides that it is in your child's be to the following reasons: The study is cancelled. | and the research team. |
| Questions, Concerns, or Complaints: If you have any questions, Concerns, or Complaints: If you have any questions research study, its procedures, risks and benefits, or should ask the Protocol Director, Dr. her at any time if you feel you have been hurt by being Independent Contact: If you are not satisfied with how have any concerns, complaints, or general questions about participant, please contact the Stanford Institutional Revindependent of the research team at also write to the Stanford IRB, Stanford University, The extra copy of this signed and dated consent form is | r alternative courses of treatment, you have a part of this study. this study is being conducted, or if you hout the research or your rights as a view Board (IRB) to speak to someone . You can |
| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g., parent, guardian or conservator) | |
| (If available) Signature of Other Parent or Guardian | Date |

Print Name of Other Parent or Guardian

The IRB determined that the permission of one parent is sufficient in accordance with 45 CFR 46.408(b).

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

| FOR QUESTIONS ABOUT THE STUDY, | <b>CONTACT:</b> | Dr. | , at |
|--------------------------------|-----------------|----------|------|
| | , or by | phone at | |

**DESCRIPTION:** Your child is invited to participate in a research study on how promoting drinking water in schools impacts what students eat and drink throughout the school day, and also their growth.

Drinking water can help children learn, maintain healthy weight, and prevent cavities. Yet at many schools, students have limited access to water during the school day.

Your child's school principal has agreed to allow researchers to conduct evaluation activities to understand how the project impacts what students eat and drink and also their growth. Your child will be asked to:

- Allow researchers to visit the school to observe what students drink at school.
- Allow Dr. and her research team to complete height and weight measurements. Dr. and her research team will use standard techniques outlined by the National Health and Nutrition Examination Survey Anthropometry Procedures Manual. Height and weight measurements are similar to how your child is measured at the doctor's office and in schools in 5th, 7th, and 9th grade. Measurements of students will occur one at a time and will take place in a private area. Students will only be asked to remove heavy coats and shoes for the measurements. We will take these measurements three times -- once now, once again before the end of the school year and once more during the next school year.
- Participate in short surveys. At the same time as the height and weight measurements, your child will be asked to complete a short survey with questions about beverage intake, screen time, and physical activity.
- Complete food and beverage diaries. Researchers will teach your child's class how to fill out a 24-hour diary to record all the food and beverages they consume in one day. Your child will be asked to complete the diary at home with your help two times -- once now and once again before the end of the school year.

The National Institutes of Health is providing financial support and/or material for this study.

**RISKS AND BENEFITS:** The risks associated with this study are minimal and include the possibility (1) that your child may feel uncomfortable while being measured and weighed and (2) loss of privacy. We will ensure that all height and weight measurements are collected quietly and in a private area. We will also do our best to protect the information we collect from your child. Information that identifies your child will be kept secure. The height and weight measurements and food and beverage diaries will not include details that directly identify your child, such as your child's name or address. Only a small number of researchers will have direct access to the information. Any reports from the study will not mention individual children or schools.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

Another possible risk is that underweight children could lose weight as a result of this study. If your child is considered to be underweight (their Body Mass Index or BMI is in the fifth percentile or lower), Dr. will contact you to discuss strategies for healthy weight management.

We cannot and do not guarantee or promise that your child will receive any benefits from this study. However, the information that your child provides may help schools, public health officials, policymakers to better understand how improvements in water access and promotion affects what students eat and drink, and their health. Your child is free to not participate in the study. If you decide not to allow your child to take part in this study, there will be no penalty to you or your child, and your child's relationship with his/her school or Stanford University will not be impacted in any way.

**TIME INVOLVEMENT:** Your child's participation in this study will take approximately 2.5 hours total over the course of the 18 month study.

**PAYMENTS:** Your child will receive a \$10 movie theater gift card after turning in all food and beverage diaries and surveys for his/her participation.

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to allow your child to participate in this project, please understand your child's participation is voluntary and you have the right to withdraw your consent or discontinue your child's participation at any time without penalty or loss of benefits to which you are otherwise entitled. The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your child's identity will not be disclosed. Your child has the right to refuse to answer particular questions.

CERTIFICATE OF CONFIDENTIALITY: This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

It is possible that, based on information gained from this study, the researchers may have serious concerns (relating to matters such as severe depression, physical abuse, etc.) about your child's health and/or safety; in such a case, the researchers may contact you and provide a referral for your child's care. It is possible that, based on information gained from this study,

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

the researchers may be required to report information (e.g., information relating to suicide, physical or sexual abuse) to the appropriate authorities.

IRB Use Only Approval Date: July 31, 2019

Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## **Authorization To Use Your Child's Health Information** For Research Purposes

Because information about your child and your child's health is personal and private, it generally cannot be used in this research study without your written authorization. If you sign this form, it will provide that authorization. The form is intended to inform you about how your child's health information will be used or disclosed in the study. Your child's information will only be used in accordance with this authorization form and the informed consent form and as required or allowed by law. Please read it carefully before signing it.

## What is the purpose of this research study and how will my child's health information be utilized in the study?

This is a research study to investigate how promoting drinking water in schools impacts what students eat and drink, and their growth. The information that your child provides may help schools, public health officials, and policymakers to better understand how promoting water in schools can affect students' health. The results of this research study may be presented at scientific meetings, published in scientific journals, or provided in reports to the funding agency, the National Institutes of Health. However, your child's identity and your child's school name will not be disclosed.

## Do I have to sign this authorization form?

You do not have to sign this authorization form. But if you do not, your child will not be able to participate in this research study. Signing the form is not a condition for receiving any medical care outside of the study.

## If I sign, can I revoke it or withdraw from the research later?

If you allow your child to participate, you are free to withdraw your authorization regarding the use and disclosure of your child's health information (and to discontinue any other participation in the study) at any time. After any revocation, your child's health information will no longer be used or disclosed in the study, except to the extent that the law allows us to continue using your child's information (e.g., necessary to maintain integrity of research). If you wish to revoke your authorization for the research use or disclosure of your child's health information in this study, you must write to:

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: <u>July 31, 2020</u>

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## What Personal Information Will Be Obtained, Used or Disclosed?

Your child's health information related to this study name, date of birth, height/weight, and beverage and food intake may be used or disclosed in connection with this research study.

## Who May Use or Disclose the Information?

The following parties are authorized to use and/or disclose your child's health information in connection with this research study:

- The Protocol Director, Dr.
- The Stanford University Administrative Panel on Human Subjects in Medical Research and any other unit of Stanford University as necessary
- Research Staff

## Who May Receive or Use the Information?

The parties listed in the preceding paragraph may disclose your child's health information to the following persons and organizations for their use in connection with this research study:

- The Office for Human Research Protections in the U.S. Department of Health and Human Services
- National Institutes of Health

Your child's information may be re-disclosed by the recipients described above, if they are not required by law to protect the privacy of the information.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

| Protocol Director: |
|---------------------|
| Projector infector |
| i iotocci Biioctoi. |

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## When will my authorization expire?

Your authorization for the use and/or disclosure of your child's health information will end on May 31, 2030 or when the research project ends, whichever is earlier.

| Signature of Legally Authorized Representative (LAR) (e.g., parent, guardian or conservator) | Date |
|---|---|
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g., parent, quardian or conservator) | |

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director: Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and

| Obesity | ess and i formation on Beverage induce and |
|---|---|
| and the research team may also withdraw consent for one or more of the following reasons: Failure to follow the instructions of decides that it is in your child the study is cancelled. | and the research team. |
| Questions, Concerns, or Complaints: If you have an this research study, its procedures, risks and benefit should ask the Protocol Director, her at any time if you feel you have been hurt by be Independent Contact: If you are not satisfied with have any concerns, complaints, or general questions participant, please contact the Stanford Institutional independent of the research team at also write to the Stanford IRB, Stanford University, The extra copy of this signed and dated consent for | ts, or alternative courses of treatment, you have a part of this study. How this study is being conducted, or if you have about the research or your rights as a likeview Board (IRB) to speak to someone have a conducted. You can |
| Signature of Legally Authorized Representative (LAF (e.g., parent, guardian or conservator) | R) Date |
| Print Name of LAR | |
| LAR's Authority to Act for Participant (e.g., parent, guardian or conservator) | |
| (If available) Signature of Other Parent or Guardian | <br>Date |
| Print Name of Other Parent or Guardian | |

The IRB determined that the permission of one parent is sufficient in accordance with 45 CFR 46.408(b).

#### Assent

(For ages 17 and under)

Approval Date: August 20, 2018

**Study Title:** Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

#### 1. What will happen to me in this study?

This is a research study about what students drink. Dr. from the Stanford University Department of Pediatrics is doing this study to learn more about how having cold and appealing water in schools changes what students eat and drink during the day, and also how it affects their growth.

Your parents were asked to give their permission for you to be in this study. If you are filling out this form, your parents have agreed for you to be in the study.

If your parents agree for you to participate in the study, and you want to participate, here's what will happen:

- Researchers will teach you how to fill out a diary to record everything you eat and drink for one day. You will fill out the diary at home with your parents two times.
- Researchers will also ask you questions about the different drinks you drink and how much time you spend watching TV and being active.
- Researchers will come to your class to weigh you and measure your height three times. They will do this quietly in a private area away from other students.

#### 2. Can anything bad happen to me?

There is a small possibility that you could lose weight during this this study. If you are at an unhealthy weight, we will talk with your parents about your weight. You are free to stop participating in the study at any time if you do not like it.

It is possible that researchers may learn information from this study that may make them concerned about your health and/or safety; in such a case, the researchers may tell your parents or someone else about it. It is possible that, based on information gained from this study, the researchers may be required to report information (e.g., information relating to suicide, physical or sexual abuse) to the appropriate authorities.

#### 3. Can anything good happen to me?

If you take part in the study, you will receive a \$10 gift card after the last time you fill out surveys.

### 4. Who can I talk to about the study?

| If you have any questions about t | ne study or any problems | s to do with | the study | you can |
|---|---|---|---|---|
| contact the Protocol Director, Dr. | . You can call | l her at | | |

the study, you can call the Stanford Institutional Review Board (IRB) at

If you have questions about the study but want to talk to someone else who is not a part of

su\_assent rev 01/07/15 

#### **Assent**

(For ages 17 and under)

#### 5. Will anyone know I am in the study?

Your participation in the study will be kept secret. The only people who will know your responses and information will be the members of the research team.

#### 6. What happens if I get hurt?

Nothing you do in this study will hurt you.

#### 7. What if I do not want to do this?

If your parents agree, you can be in the study if you want to. But you don't have to be in it if you don't want to. Nobody will get mad at you if you don't want to do this.

If you decide to be in the study now and you change your mind later, that's okay. You just have to tell the study researchers as soon as you change your mind, and you will be taken out of the study.

## SIGNATURE

| If you agree to be in this study, please sign here: | |
|-----------------------------------------------------|------|
| Signature of Child | Date |
| Printed name of Child | |

su\_assent rev 01/07/15 

#### Assent

(For ages 17 and under)

Approval Date: August 20, 2018

**Study Title:** Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

#### 1. What will happen to me in this study?

This is a research study about what students drink. Dr. from the Stanford University Department of Pediatrics is doing this study to learn more how to change the drinks that students drink during the day.

New reusable water bottle filling stations will be installed at your school. There will also be signs about drinks posted in different places at the school. All the students in your class will receive a reusable water bottle to leave overnight at school and another one to take home. Students will fill up their water bottles every morning, and keep their water bottles on or near their desks to drink from during class. Also, researchers will come to your class eight times to teach short lessons about why it is important to drink water. They will give you also give you short fun activities to complete at home. You will also get prizes during the classes.

Your parents were asked to give their permission for you to be in this study. If you are filling out this form, your parents have agreed for you to be in the study.

If your parents agree for you to participate in the study, and you want to participate, here's what will happen:

- Researchers will teach you how to fill out a diary to record everything you eat and drink for one day. You will fill out the diary at home with your parents two times.
- Researchers will also ask you questions about the different drinks you drink and how much time you spend watching TV and being active.
- Researchers will come to your class to weigh you and measure your height three times. They will do this quietly in a private area away from other students.

#### 2. Can anything bad happen to me?

There is a small possibility that you could lose weight during this this study. If you are at an unhealthy weight, we will talk with your parents about your weight. You are free to stop participating in the study at any time if you do not like it.

It is possible that researchers may learn information from this study that may make them concerned about your health and/or safety; in such a case, the researchers may tell your parents or someone else about it. It is possible that, based on information gained from this study, the researchers may be required to report information (e.g., information relating to suicide, physical or sexual abuse) to the appropriate authorities.

#### 3. Can anything good happen to me?

If you take part in the study, you will receive a \$10 movie ticket gift card after the last time you fill out surveys.

su\_assent rev 01/07/15 

Assent
(For ages 17 and under)

| 4. | Who can I talk to about the study? If you have any questions about the study or any problems to do with the study you can contact the Protocol Director, Dr. You can call her at |
|---|---|
| | If you have questions about the study but want to talk to someone else who is not a part of the study, you can call the Stanford Institutional Review Board (IRB) at |
| 5. | Will anyone know I am in the study? Your participation in the study will be kept secret. The only people who will know your responses and information will be the members of the research team. |
| 6. | What happens if I get hurt? Nothing you do in this study will hurt you. |
| 7. | What if I do not want to do this? If your parents agree, you can be in the study if you want to. But you don't have to be in it if you don't want to. Nobody will get mad at you if you don't want to do this. |
| | If you decide to be in the study now and you change your mind later, that's okay. You just have to tell the study researchers as soon as you change your mind, and you will be taken out of the study. |
| | SIGNATURE |
| | If you agree to be in this study, please sign here: |
| | Signature of Child Date |

 su\_assent rev 01/07/15

Printed name of Child

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

### FOR QUESTIONS ABOUT THE STUDY, CONTACT: Dr.

, at

**DESCRIPTION:** You are invited to participate in a research study on how improving access to drinking water and promoting the consumption of drinking water impacts what students drink throughout the school day.

Drinking water can help children learn and can help them maintain a healthy weight and teeth. Yet at many schools, students have limited access to water during the school day. The primary goal of our study is to examine the impact of installing new water stations and promoting water consumption. Results from this study will be used to develop programs and policies to encourage students to consume water at school.

In order to help us understand if there are any programs, other than the water program, that could affect what students at your school eat or drink or their weight, you will be asked to complete a hand-written survey about nutrition and physical activity policies and practices at your school. The survey should take about 20 minutes to complete. We will ask you to complete the survey two times -- once now and once again before the end of the study.

**RISKS AND BENEFITS:** The risks associated with this study are minimal and include the possibility that you may not want to answer some of the questions on the surveys because they make you uncomfortable. You are free to decline to answer any questions you do not wish to answer. We will do our best to protect the information we collect from you. Information that identifies you and your school will be kept secure. The surveys will not include details that directly identify you or your school, such as your name or address. The information gathered will be kept secure and separate from information that identifies you. Only a small number of researchers will have direct access to the information. If the study is published or presented at scientific meetings, names and other information that might identify you will not be used. No reports from this research will be provided to state agencies and specific individuals will not be identified in any study information that is published or presented at conferences.

We cannot and do not guarantee or promise that you will receive any benefits from this study. However, the information that you provide may help public health officials, policymakers, and facility staff to better understand how to improve access to healthy beverages for kids at school. Your decision whether or not to participate in this study will not affect your employment/medical care.

**TIME INVOLVEMENT:** Your participation in this experiment will take approximately 40 minutes total over the course of 15 months.

**PAYMENTS:** You will receive a \$50 gift card after the last time you fill out the survey as payment for your participation.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to participate in this project, please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your identity will not be disclosed. You have the right to refuse to answer particular questions.

#### WITHDRAWAL FROM STUDY:

The Protocol Director may also withdraw you from the study, without your consent for one or more of the following reasons:

- o Failure to follow the instructions of Dr. and the research team.
- The study is cancelled.

#### **CERTIFICATE OF CONFIDENTIALITY:**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

#### **CONTACT INFORMATION:**

| Questions, Concerns, or Complaints: If you have any | y questions, concerns or complaints about |
|---|---|
| this research study, its procedures, risks and benefit | s, or alternative courses of treatment, you |
| should ask the Protocol Director, | . You should also contact |
| her at any time if you feel you have been hurt by be | ing a part of this study. |

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at also write to the Stanford IRB, Stanford University,

*IRB Use Only*Approval Date: July 31, 2019
Expiration Date: <u>July 31, 2020</u>

| Donata and Discostant |
|-----------------------|
| Protocol Director: |

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

| The extra copy of this signed and dated conse | nt form is for you to keep. |
|-----------------------------------------------|-----------------------------|
| Signature of Adult Participant | Date |
| Print Name of Adult Participant | |

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

Protocol Director:

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

## FOR QUESTIONS ABOUT THE STUDY, CONTACT: Dr.

, or by phone at (

**DESCRIPTION:** You are invited to participate in a research study on how improving access to drinking water and promoting the consumption of drinking water impacts what students drink throughout the school day.

Drinking water can help children learn and can help them maintain a healthy weight and teeth. Yet at many schools, students have limited access to water during the school day. The primary goal of our study is to examine the impact of installing new water stations and promoting water consumption. Results from this study will be used to develop programs and policies to encourage students to consume water at school.

In order to help us understand if there are any programs, other than the water program, that could affect what students at your school eat or drink or their weight, you will be asked to complete an online or paper survey about nutrition and physical activity policies and practices at your school. The survey should take about 20 minutes to complete. We will ask you to complete the survey two times -- once now and once again before the end of the study.

**RISKS AND BENEFITS:** The risks associated with this study are minimal and include the possibility that you may not want to answer some of the questions on the surveys because they make you uncomfortable. You are free to decline to answer any questions you do not wish to answer. We will do our best to protect the information we collect from you. Information that identifies you and your school will be kept secure. The surveys will not include details that directly identify you or your school, such as your name or address. The information gathered will be kept secure and separate from information that identifies you. Only a small number of researchers will have direct access to the information. If the study is published or presented at scientific meetings, names and other information that might identify you will not be used. No reports from this research will be provided to state agencies and specific individuals will not be identified in any study information that is published or presented at conferences.

We cannot and do not guarantee or promise that you will receive any benefits from this study. However, the information that you provide may help public health officials, policymakers, and facility staff to better understand how to improve access to healthy beverages for kids at school. Your decision whether or not to participate in this study will not affect your employment/medical care.

**TIME INVOLVEMENT:** Your participation in this experiment will take approximately 40 minutes total over the course of 15 months.

**PAYMENTS:** You will receive a \$50 gift card after the last time you fill out the survey as payment for your participation.

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

| Protocol Director: |
|--------------------|
| ETOIOCOLEMECIOL |

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

**PARTICIPANT'S RIGHTS:** If you have read this form and have decided to participate in this project, please understand your participation is voluntary and you have the right to withdraw your consent or discontinue participation at any time without penalty or loss of benefits to which you are otherwise entitled. The results of this research study may be presented at scientific or professional meetings or published in scientific journals. However, your identity will not be disclosed. You have the right to refuse to answer particular questions.

#### WITHDRAWAL FROM STUDY:

The Protocol Director may also withdraw you from the study, without your consent for one or more of the following reasons:

- o Failure to follow the instructions of Dr. and the research team.
- The study is cancelled.

#### **CERTIFICATE OF CONFIDENTIALITY:**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers with this Certificate may not disclose or use information, documents, or biospecimens that may identify you in any federal, state, or local civil, criminal, administrative, legislative, or other action, suit, or proceeding, or be used as evidence, for example, if there is a court subpoena, unless you have consented for this use. Information, documents, or biospecimens protected by this Certificate cannot be disclosed to anyone else who is not connected with the research except, if there is a federal, state, or local law that requires disclosure (such as to report child abuse or communicable diseases but not for federal, state, or local civil, criminal, administrative, legislative, or other proceedings, see below); if you have consented to the disclosure, including for your medical treatment; or if it is used for other scientific research, as allowed by federal regulations protecting research subjects.

#### **CONTACT INFORMATION:**

| Questions, Concerns, or Complaints: If you have any questions, cor | ncerns or complaints about |
|---|---|
| this research study, its procedures, risks and benefits, or alternative | e courses of treatment, you |
| should ask the Protocol Director, Dr. | . You should also contact |
| her at any time if you feel you have been hurt by being a part of th | is study. |

Independent Contact: If you are not satisfied with how this study is being conducted, or if you have any concerns, complaints, or general questions about the research or your rights as a participant, please contact the Stanford Institutional Review Board (IRB) to speak to someone independent of the research team at also write to the Stanford IRB, Stanford University,

IRB Use Only
Approval Date: July 31, 2019
Expiration Date: July 31, 2020

| I |
|---------------------|
| Protocol Director: |
| Prolocol Director |
| ii iotocoi biiotoi. |

Protocol Title: Water First: The Impact of School Water Access and Promotion on Beverage Intake and Obesity

| The extra copy of this signed and dated consen | t form is for you to keep. |
|------------------------------------------------|----------------------------|
| Signature of Adult Participant | <br>Date |
| Print Name of Adult Participant | |